CLINICAL TRIAL: NCT02157064
Title: Autologous Adipose Stromal Vascular Fraction Outcomes Research Study
Brief Title: Outcomes Data of Adipose Stem Cells to Treat Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: StemGenex (Industry)
Responsible Party: Sponsor
Other Study IDs: SVF01MS; ASCMS-01 (Other: StemGenex)
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the impact that treatment with a cellular concentrate derived from an individual's own fat, known as the stromal vascular fraction (SVF), has on the quality of life of people with multiple sclerosis (MS). SVF contains components with "regenerative" properties, including stem cells that may be capable of ameliorating specific disease conditions. This study is designed to evaluate quality of life changes in individuals with MS for up to 12 months following SVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for a stem cell/SVF treatment
* Subjects diagnosed with some form of multiple sclerosis
* Subjects between the ages of 18 and 65
* Subjects willing and able to sign informed consent
* Subjects willing and able to perform follow up interviews and surveys

Exclusion Criteria:

* Subjects for whom baseline data is not available
* Subjects with additional major health diagnoses
* Subjects that are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2014-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Quality of Life Over the Course of a 12 Month Period as Measured by the Multiple Sclerosis Quality of Life Inventory (MSQLI) | Baseline, 12 months
  The change from baseline over the course of 12 months using participants' assessment of their quality of life. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 3, 6, and 12). Answer options are graded on a multiple point Likert scale.

SECONDARY OUTCOMES:
Change from Baseline in Overall General Quality of Life Over the Course of a 12 Month Period as Measured by the Health Status Questionnaire (SF-36) | Baseline, Month 12
  Change from Baseline in General Quality of Life at Month 12 as Measured by Participants Using the Health Status Questionnarie (SF-36)
Change from Baseline in Fatigue Over the Course of a 12 Month Period as Measured by the Modified Fatigue Impact Scale (MFIS) | Baseline, Month 12
  Change from Baseline in Fatigue at Month 12 as Measured by Participants Using the Modified Fatigue Impact Scale (MFIS)
Change from Baseline in Pain and Other Sensory Symptoms Over the Course of a 12 Month Period as Measured by the MOS Pain Effects Scale (PES) | Baseline, Month 12
  Change from Baseline in Pain and Other Sensory Symptoms at Month 12 as Measured by Participants Using the MOS Pain Effects Scale (PES)
Change from Baseline in Sexual Satisfaction Over the Course of a 12 Month Period as Measured by the Sexual Satisfaction Scale (SSS) | Baseline, Month 12
  Change from Baseline in Sexual Satisfaction at Month 12 as Measured by Participants Using the Sexual Satisfaction Scale (SSS)
Change from Baseline in Bladder Control Over the Course of a 12 Month Period as Measured by the Bladder Control Scale (BLCS) | Baseline, Month 12
  Change from Baseline in Bladder Control at Month 12 as Measured by Participants Using the Bladder Control Scale (BLCS)
Change from Baseline in Bowel Control Over the Course of a 12 Month Period as Measured by the Bowel Control Scale (BWCS) | Baseline, Month 12
  Change from Baseline in Bowel Control at Month 12 as Measured by Participants Using the Bowel Control Scale (BWCS)
Change from Baseline in Visual Problems Over the Course of a 12 Month Period as Measured by the Impact of Visual Impairment Scale (IVIS) | Baseline, Month 12
  Change from Baseline in Visual Problems at Month 12 as Measured by Participants Using the Impact of Visual Impairment Scale (IVIS)
Change from Baseline in Cognitive Problems Over the Course of a 12 Month Period as Measured by the Perceived Deficits Questionnaire (PDQ) | Baseline, Month 12
  Change from Baseline in Cognitive Problems at Month 12 as Measured by Participants Using the Perceived Deficits Questionnaire (PDQ)
Change from Baseline in Emotional Distress Over the Course of a 12 Month Period as Measured by the Mental Health Inventory (MHI) | Baseline, Month 12
  Change from Baseline in Emotional Distress at Month 12 as Measured by Participants Using the Mental Health Inventory (MHI)
Change from Baseline in Social Support Over the Course of a 12 Month Period as Measured by the Modified MOS Social Support Survey (MSSS) | Baseline, Month 12
  Change from Baseline in Social Support at Month 12 as Measured by Participants Using the Modified MOS Social Support Survey (MSSS)

CONTACTS AND LOCATIONS:
Locations (1):
- StemGenex, San Diego, California, United States